CLINICAL TRIAL: NCT06023290
Title: Validation of Digital Heart Rhythm Devices in the Detection of Atrial Fibrillation
Acronym: VALIDATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Z-2023023
Record Dates: First submitted 2023-07-04; First posted 2023-09-05 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study population (single arm) (Other)
  Interventions: Diagnostic Test: Heart rhythm measurements with Preventicus®; Diagnostic Test: Heart rhythm measurements with FibriCheck®; Diagnostic Test: Heart rhythm measurements with Apple Watch®; Diagnostic Test: Heart rhythm measurements with 6L Kardia Mobile®

INTERVENTIONS:
Diagnostic Test: Heart rhythm measurements with Preventicus® — The sequence of the digital heart rhythm measurements is randomly assigned for each patient. The reference heart rhythm is determined by a simultaneous recording with a 12-lead ECG as gold standard.
Diagnostic Test: Heart rhythm measurements with FibriCheck® — The sequence of the digital heart rhythm measurements is randomly assigned for each patient. The reference heart rhythm is determined by a simultaneous recording with a 12-lead ECG as gold standard.
Diagnostic Test: Heart rhythm measurements with Apple Watch® — The sequence of the digital heart rhythm measurements is randomly assigned for each patient. The reference heart rhythm is determined by a simultaneous recording with a 12-lead ECG as gold standard.
Diagnostic Test: Heart rhythm measurements with 6L Kardia Mobile® — The sequence of the digital heart rhythm measurements is randomly assigned for each patient. The reference heart rhythm is determined by a simultaneous recording with a 12-lead ECG as gold standard.

SUMMARY:
The VALIDATION study aims to evaluate the performance of four state-of-the-art digital heart rhythm devices (Preventicus®, FibriCheck®, Apple Watch®, 6L Kardia Mobile®) for the detection of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* The patient is an ambulatory cardiology patient.
* The patient is at least 18 years old.
* The patient is sinus or in atrial fibrillation.
* The patient is able to perform the study procedures together with the study assistant.

Exclusion Criteria:

* Patients with a pacemaker
* Inclusion in another clinical trial that may influence the results of this trial
* The patient is unable to comprehend the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Sensitivity | During the heart rhythm measurements
  Proportion of true positives tests with the device of interest out of all patients with AF on the 12-lead ECG.
Specificity | During the heart rhythm measurements
  Proportion of true negative tests with the device of interest out of all patients in sinus rhythm on the 12-lead ECG.
Accuracy | During the heart rhythm measurements
  Proportion of correct classifications with the device of interest. Correct classification is provided by the 12-lead ECG.
Cramer's V | During the heart rhythm measurements
  The association of between the classification by the device of interest versus the 12-lead ECG, expressed as Cramer's V.

SECONDARY OUTCOMES:
Positive predictive value | During the heart rhythm measurements
  Proportion of true positive tests out of all positive tests.
Negative predictive value | During the heart rhythm measurements
  Proportion of true negative tests out of all negative tests.
Patient preference score (for the use of the diagnostic devices) | During the heart rhythm measurements
  This score is a (1-5) ordinal result based on the VALIDATION study questionnaire.

OTHER OUTCOMES:
Sensitivity, specificity and Cramer's V using only measurements of sufficient quality for analysis | During the heart rhythm measurements
  The proportion of true positive tests, true negative tests and the association of between the classification of the test devices and 12-lead ECG.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium